CLINICAL TRIAL: NCT03606694
Title: Effect of Dihydromirycetin Administration on Glycemic Control, Insulin Sensitivity and Insulin Secretion in Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of Dihydromirycetin on Glycemic Control, Insulin Sensitivity and Insulin Secretion in Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Karina Griselda Pérez Rubio, Principal Investigator, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DHM-Metformin-T2DM
Record Dates: First submitted 2018-07-20; First posted 2018-07-31 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: dihydromyricetin; metformin; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dihydromyricetin; Metformin

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dihydromyricetin (Experimental): Dihydromyricetin capsules, 300 mg, two times per day before break-fast and dinner during 12 weeks.
  Interventions: Drug: Dihydromyricetin
- Metformin (Experimental): Metformin capsules, 850 mg, two times per day before break-fast and dinner during 12 weeks.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Dihydromyricetin — The intervention wiil be 300 mg, two times per day before break-fast and dinner during 12 weeks.
  Other Names: Ampelopsis grossedentata Extract
  Arms: Dihydromyricetin
Drug: Metformin — The intervention wiil be 850 mg, two times per day before break-fast and dinner during 12 weeks.
  Other Names: Brad Predial
  Arms: Metformin

SUMMARY:
Dihydromyricetin has demonstrated promising effects in glycemic control, insulin sensitivity and insulin secretion, that above mentioned findings show that dihydromyricetin has an excellent potential effect in the treatment of type 2 diabetes mellitus patients.

DETAILED DESCRIPTION:
A double-blind, randomized clinical trial of three pharmacological groups in 36 patients with a diagnosis of type 2 diabetes mellitus in accordance with the American Diabetes Association (ADA) without treatment.

They will be assigned randomly two groups of 12 patients, each one will receive dihydromyricetin 300 mg or metformin 850 mg, two times per day before having break-fast and before having dinner during 12 weeks.

The Area Under the Curve of glucose and insulin will be calculated, total insulin secretion (Insulinogenic index), first-phase of insulin secretion (Stumvoll index) and insulin sensitivity (Matsuda index).

This protocol is already approved by the local ethics committee and written informed consent it's going to be obtained from all volunteers.

Statistical analysis will be presented through measures of central tendency and dispersion, average and deviation standard for quantitative variables; frequencies and percentages for variable qualitative. Qualitative variables will be analyzed by X2, will be used for differences inter-group Mann-Whitney U Test and Wilcoxon Test for the within-groups differences. It will be considered statistical significance p ≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients both sexes
* Age between 30 and 60 years
* Diabetes mellitus type 2 of recent diagnosis without pharmacological treatment, with one of the following criteria (fasting blood glucose levels >126 mg/dL; postprandial blood glucose levels after an oral glucose tolerance test with 75 of oral glucose >200 mg/dl; or glycosylated hemoglobin between >6.5%)
* Informed consent signed

Exclusion Criteria:

* Women with confirmed or suspected pregnancy, or under lactation and/or puerperium
* Previous treatment for glucose
* Fasting glucose ≥250 mg/dL
* Body Mass Index ≥34.9 kg/m2
* Known uncontrolled renal, hepatic, heart or thyroid diseased
* Hypersensibility to ingredients of intervention
* Triglycerides ≥500 mg/dL
* Total cholesterol ≥240 mg/dL
* Blood Pressure ≥140/90 mmHg

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Fasting glucose | Baseline to Week 12
  Changes in fasting glucose levels after 12 weeks of intervention with dihydromyricetin and metformin. The fasting glucose levels will be evaluated at baseline and week 12 with enzymatic/colorimetric techniques and the entered values reflect the fasting glucose level at week 12.
Postprandial glucose | Baseline to Week 12
  Changes in postprandial glucose levels after 12 weeks of intervention with dihydromyricetin and metformin. Postprandial glucose will be evaluated at baseline and week 12 after a oral glucose tolerance test with enzymatic/colorimetric techniques and the entered values reflect the insulin sensitivity at week 12.
Glycosylated hemoglobin | Baseline to Week 12
  Changes in glycosylated hemoglobin (A1C) after 12 weeks of intervention with dihydromyricetin and metformin. Glycosylated hemoglobin will be evaluated at baseline and week 12 by high pressure liquid chromatography (HPLC) and the entered values reflect the glycosylated hemoglobin at week 12.
Insulin sensitivity | Baseline to Week 12
  Insulin sensitivity will be calculated at baseline and week 12 with Matsuda index and the entered values reflect the insulin sensitivity at week 12.
Total insulin secretion | Baseline to Week 12
  Total insulin secretion will be calculated at baseline and week 12 with insulinogenic index and the entered values reflect the total insulin secretion at week 12.
First phase of insulin secretion | Baseline to Week 12
  The first phase of insulin secretion will be calculated at baseline and week 12 with Stumvoll index and the entered values reflect the first phase of insulin secretion at week 12.

SECONDARY OUTCOMES:
Waist Circumference | Baseline to Week 12
  Waist circumference will be evaluated at baseline and at week 12 with a flexible tape.
Body Weigh | Baseline, week 4, week 8 and week 12
  The body weight will be measured at baseline, week 4, week 8 and week 12 with a bioimpedance balance and the entered values reflect the body weight at week 12.
Body Mass Index | Baseline, week 4, week 8 and week 12
  Body Mas Index will be calculated at baseline, week 4, week 8 and week 12 with the Quetelet index formula and the entered values reflect the body mass index at week 12.
C reactive protein | Baseline to Week 12
  C reactive protein will be evaluated at baseline and week 12 by enzyme-linked immunosorbent assay (ELISA) and the entered values reflect the creatinine levels at week 12
Interleukin 6 | Baseline to Week 12
  Interleukin 6 will be evaluated at the beginning and during week 12 using the enzyme-linked immunosorbent assay (ELISA) and the values entered reflect creatinine levels at week 12
Total Cholesterol | Baseline to Week 12
  Total cholesterol levels will be evaluated at baseline and week 12 by enzymatic/colorimetric techniques and the entered values reflect the total cholesterol level at week 12
Triglycerides levels | Baseline to Week 12
  Triglycerides levels will be evaluated at baseline and week 12 with enzymatic/colorimetric techniques and the entered values reflect the triglycerides level at week 12
High Density Lipoprotein (c-HDL) levels | Basline to Week 12
  c-HDL levels will be evaluated at baseline and week 12 with enzymatic/colorimetric techniques and the entered values reflect the c-HDL level at week 12
Low Density Lipoproteins (c-LDL) levels | Baseline to Week 12
  c-LDL levels will be evaluated at baseline and week 12 with enzymatic/colorimetric techniques and the entered values reflect the c-LDL level at week 12
Creatinine levels | Baseline to Week 12
  Creatinine levels will be evaluated at baseline and week 12 with enzymatic/colorimetric techniques
Alanine aminotransferase (ALT) levels | Baseline to Week 12
  ALT levels will be evaluated at baseline and week 12 with enzymatic/colorimetric techniques
Aspartate aminotransferase (AST) levels | Baseline to Week 12
  AST levels will be evaluated at baseline and week 12 with enzymatic/colorimetric techniques
Blood pressure | Baseline to Week 12
  Blood pressure will be measured at baseline and week 12 with a digital sphygmomanometer and the entered values reflect the blood pressure at week 12

CONTACTS AND LOCATIONS:
Overall Officials: MANUEL GONZALEZ ORTIZ, PhD, Principal Investigator — Instituto de Terapeútica Experimental y Clínica. Universidad de Guadalajara
Locations (1):
- Instituto de Terapeútica Experimental y Clínica. Centro Universitario de Ciencias de la Salud. Universidad de Guadalajara, Guadalajara, Jalisco, Mexico